CLINICAL TRIAL: NCT05762146
Title: Networked Drug REpurposing for Mechanism-based neuroPrOtection in Ischaemic STROKE (REPO-STROKE IIa)
Brief Title: Networked Drug REpurposing for Mechanism-based neuroPrOtection in Acute Ischaemic STROKE
Acronym: REPO-STROKE II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REPO-STROKE II; 2019-000474-31 (EudraCT Number)
Record Dates: First submitted 2022-08-23; First posted 2023-03-09 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke | interventions — riociguat; Propylthiouracil; Perphenazine

STUDY DESIGN:
Intervention Model Description: This is a Prospective Randomized Open-label Blinded End-point (PROBE) trial evaluating safety and efficacy of a triple combination therapy of riociguat, propylthiouracil, and perphenazine, administered orally in addition to standard of care treatment in patients with disabling acute ischemic stroke. Patients will be randomly assigned to the triple combination therapy group or the control group in a 3:1 ratio:
Who Masked: Outcomes Assessor
Masking Description: This is a Prospective Randomized Open-label Blinded End-point (PROBE) trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Riociguat +Propylthiouracil +Perphenazine (Experimental): Triple combination therapy group:
  ○ each patient in this group will receive two doses (8 +/- 2 hours between doses) of orally administered combination therapy of riociguat, propylthiouracil, and perphenazine, in addition to standard of care.
  Interventions: Drug: Riociguat; Drug: Propylthiouracil; Drug: Perphenazine
- standard of care (No Intervention): Control group: each patient in this group will receive only standard of care

INTERVENTIONS:
Drug: Riociguat — Riociguat is an sGC stimulator currently approved and marketed for pulmonary arterial hypertension.
  Other Names: Adempas
  Arms: Riociguat +Propylthiouracil +Perphenazine
Drug: Propylthiouracil — Propylthiouracil, already marketed for the treatment of various subtypes of hyperthyroidism, has been identified as a new member of the class of potent and effective neuronal nitric oxide synthase (NOS1) inhibitors
  Other Names: Propycil
  Arms: Riociguat +Propylthiouracil +Perphenazine
Drug: Perphenazine — Perphenazine, already marketed as an antiemetic and antipsychotic drug, presents the best NADPH oxidase (NOX) inhibitory characteristics compared to other compounds of the same drug class.
  Other Names: Perphenazin neuraxpharm
  Arms: Riociguat +Propylthiouracil +Perphenazine

SUMMARY:
A combination therapy proposed to be evaluated in this trial, consisting of three already registered compounds with a validated disease mechanism and with known safety profiles, targets key proteins in the dysregulated signal network in stroke, and is expected to synergistically result in post-stroke blood-brain barrier stabilization and neuroprotection. The synergistic mode of action will allow for low doses and is expected to reduce possible side effects while maintaining maximal efficacy

DETAILED DESCRIPTION:
There is a high need for new drugs & novel approaches for neuroprotection in stroke treatment.

Pre-clinically, three interrelated in silico predicted drug targets and pharmacological principles all belonging to the same signal network were validated at the preclinical level to be causally relevant in stroke and thus hold promise for the first-in-class mechanism-based, curative neuroprotective therapy of an ischemic stroke:

1. NADPH oxidase type 4 and 5 (NOX4, NOX5), members of a reactive oxygen radical (ROS) forming enzyme family being either upregulated during hypoxia or activated by high post-reperfusion calcium influx causing unphysiological high levels of ROS and thereby blood-brain barrier (BBB) breakdown and neuronal damage, which can be prevented by NOX inhibitors (NOXi).
2. Nitric oxide (NO) synthase type 1 (NOS1), a neuronal signaling enzyme, which in stroke is hyperactivated (excitotoxicity) and produces neurotoxic quantities of NO, which are further toxified by chemically interacting with NADPH oxidase-derived ROS, forming and even more toxic peroxynitrite and which can be prevented by NOS inhibitors (NOSi)
3. Soluble guanylate cyclase (sGC), an enzyme, which forms the BBB stabilizing and neuroprotective second messenger, cyclic GMP (cGMP), but upon stroke is oxidatively damaged to a heme-free apo sGC (by peroxynitrite). Moreover, any remaining sGC is less activated by NO, because NO is scavenged by ROS and deviated into peroxynitrite. Thus, cGMP formation is greatly reduced in stroke, which can be reversed by sGC modulators which increase the activity of both sGC and apo-sGC in an NO-independent manner and thereby reinstall cGMP formation, BB closure and neuroprotection.

Different representatives of the drug classes of NADPH oxidase inhibitors (NOXi), nitric oxide synthase inhibitors (NOSi), and soluble guanylate cyclase modulators were identified and shown to be highly effective when given alone in different small animal experimentation and in vitro human models. However, since all single target approaches in stroke have so far failed in clinical development during the last decades, and NOS, NOX and sGC all belong to the same disease module, an innovative combined, so-called network pharmacology approach is proposed, i.e., a combination of 3 already registered compounds with a validated disease mechanism: the sGC activator riociguat, the NOS1 inhibitor propylthiouracil, and the NOX inhibitor perphenazine.

Riociguat is an sGC stimulator currently approved and marketed for pulmonary hypertension. Post-reperfusion therapy with riociguat, increased cGMP formation and therefore leads to direct neuroprotection and reduced infarct volume in a stroke animal model. Propylthiouracil is already marketed for the treatment of various subtypes of hyperthyroidism and has been identified as a new member of the class of potent and effective NOS1 inhibitors. Pre-clinically, post-reperfusion treatment with propylthiouracil significantly reduced infarct volume in brain ischemia mice models compared to non-treated animals (pre-clinical in-house data, unpublished). Perphenazine is already marketed as an antiemetic and antipsychotic, has the best NOX inhibitory characteristics compared to other compounds of the same drug class, and significantly reduced infarct size in acute ischemic stroke mice models.

In summary, the combination therapy proposed to be evaluated in this trial, consisting of already registered compounds with a validated disease mechanism and with known safety profiles, targets key proteins in the dysregulated signal network in stroke, and is expected to synergistically result in post-stroke blood-brain barrier stabilization and neuroprotection. The synergistic mode of action will allow for low doses and is expected to reduce possible side effects while maintaining maximal efficacy.

ELIGIBILITY:
Inclusion criteria:

* Informed consent has to be obtained from the patient or a legal representative. In case this is not feasible due to the emergency situation, an alternative informed consent procedure is allowed, according to the current legislation in Germany, as described in section 15.4 and 15.5 of this protocol.
* Male or female adult, ≥18 to ≤80 years of age. Patients older than 80 years of age may be enrolled after review of an initial safety data set obtained from younger patients as described in section 7.2.
* Disabling acute ischemic stroke with an NIHSS score of ≤12 at time of randomization.
* Treatment with IMP can be initiated within 24 hours after the onset of stroke or after last known normal.

Exclusion criteria:

* Patients receiving intravenous thrombolysis with recombinant tissue plasminogen activator (rt-PA) for the index event (i.e., the current stroke that led to screening the patient for this trial).
* Prior inability to walk or to lead an independent life, which is defined as daily need for assistance in performing activities of daily living (ADL).
* Patients who are delirious, comatose or stuporous (a score of ≥ 2 on item 1.a of the NIHSS).
* Patients undergoing mechanical thrombectomy or intra-arterial thrombolysis.
* Detection of hemorrhage on baseline CT.
* Severe dysphagia with inability to swallow and no indication for nasogastric tube as per opinion of the investigator and thus inability to administer IMP.
* Systolic blood pressure < 110 mmHg at randomization.
* Pregnant and breastfeeding patients. Females with childbearing potential must comply with using highly effective methods of contraception as defined in section 9.2.
* Reported severe ongoing hepatic impairment (Child Pugh C).
* Reported relevant ongoing renal failure with known GFR <30ml/min.
* Reported ongoing major depression.
* Reported ongoing tracheal obstruction.
* Reported ongoing pulmonary hypertension associated with idiopathic interstitial pneumonias (PHIIP)
* Reported leucopenia or agranulocytosis.
* Reported agranulocytosis during previous treatment with thiourea derivatives.
* Reported hypersensitivity to perphenazine or propylthiouracil or riociguat or any of the other excipients.
* Participation in another clinical trial within the last four weeks.
* Reported use of phosphodiesterase (PDE) inhibitors (such as sildenafil, tadalafil, vardenafil) within the last 7 days.
* Reported use of nitrates or nitric oxide donors (such as amyl nitrite) in any form including recreational drugs called 'poppers' within the last 7 days.
* Reported use of antithyroid drugs within the last 7 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
SICH as per ECASS III | 30 days
  Frequency of symptomatic intracranial hemorrhages as per ECASS III

SECONDARY OUTCOMES:
SICH as per Heidelberg Bleeding Classification | 30 days
  Frequency of symptomatic intracranial hemorrhages as per Heidelberg Bleeding Classification
SICH as per SITSMOST | 30 days
  Frequency of symptomatic intracranial hemorrhages as per SITSMOST
SICH as per NINDS | 30 days
  Frequency of symptomatic intracranial hemorrhages as per NINDS
Mortality | 30 days
  Frequency of all cause mortality
SAE | 30 days
  All (S)AEs considered related to the triple combination therapy
Duration of hospital stay | 30 days
  Time from randomization to discharge
Duration of intensive care unit (ICU) stay | 30 days
  Period during which the patient stayed at a ward with capacity for mechanical ventilation
Duration of invasive mechanical ventilation | 30 days
  in hours
Duration of non-invasive mechanical ventilation | 30 days
  in hours
Change of initial 'volume of hypoperfusion' | 5 days
  Change in "ml" of volume of hypoperfusion in initial Computed Tomography Perfusion (CTP) to final 'volume of infarct core' as assessed through follow-up Magnetic Resonance Imaging (MRI).
Change of initial 'volume of infarct core' | 5 days
  Change in "ml" of infarct core of initial Computed Tomography Perfusion (CTP) to final 'volume of infarct core' as assessed through follow-up Magnetic Resonance Imaging (MRI).
mRS | 30 days
  Shift analysis of mRS
NIHSS change | 5 days
  Change from baseline in National Institute of Health Stroke Scale (NIHSS) score

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Department of Neurology, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casas AI, Nogales C, Szepanowski RD, Elbatreek MH, Anastasi E, Sadegh S, Skelton J, Frank B, Wipat A, Baumbach J, Kleinschnitz C, Schmidt HHHW. Synergistic Network Pharmacology: Preclinical Validation and Clinical Safety in Acute Ischemic Stroke. J Am Heart Assoc. 2025 May 20;14(10):e039098. doi: 10.1161/JAHA.124.039098. Epub 2025 May 15. PMID 40371623